CLINICAL TRIAL: NCT04585243
Title: HPV Self-sampling Among Women at the Penn State Hershey Colposcopy Clinics
Brief Title: Self-sampling for Human Papillomavirus (HPV) Among Patients Receiving Colposcopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment, preliminary analyses indicates that primary endpoint has been met
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer L. Moss, PhD, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13464
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: HPV
Keywords: HPV; Self-Sampling; Colposcopy; Cervical cancer; Cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants who enroll in the study will be asked to complete an HPV self-sampling kit in addition to completing their colposcopy exam. Participants will collect the sample at home before or after their exam and mail it back to the Penn State Health laboratory for analysis. The results will be compared to those of the clinician-collected (standard of care) colposcopy exam, Pap, and HPV test. Participants will also complete a follow up survey over the phone after their sample is collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Self-Sampling Kit (Experimental): Participants will be mailed a Self-Sampling kit (Evalyn Brush) to collect samples for analysis for HPV/Cervical cancer screening.
  Interventions: Device: Evalyn Brush

INTERVENTIONS:
Device: Evalyn Brush — The Evalyn Brush is a self-sampling kit that can be used to collect a sample to screen for HPV/Cervical cancer at home.

SUMMARY:
This study seeks to compare the accuracy and acceptability of HPV testing self-sampling kit and standard clinician-sampling for HPV testing. The primary outcome of this study is the concordance between screening results on self-sampling kits compared to clinician-collected HPV test, Pap smear results, and colposcopy. Secondary endpoints will include acceptability of self-sampling and barriers to cervical cancer screening. These endpoints will be analyzed to try to circumvent barriers to the cervical cancer screening and ascertain whether self-sampling is a viable alternative.

DETAILED DESCRIPTION:
The American Cancer Society estimates that 4,170 women in the United States (US) will die from cervical cancer in 2018 (Siegel et al., 2018). Screening can reduce cancer mortality by (1) detecting malignancies when they are more treatable and (2) for some tests, identifying precancerous lesions for removal (Shieh et al., 2016). Guidelines recommend cytology and/or HPV testing for cervical cancer screening among women ages 30-65 years, but screening rates are suboptimal (U.S. Preventive Services Task Force, 2018; Saslow et al., 2012).

To help bridge these gaps in screening, HPV self-sampling would be an alternative to clinical-sampling for HPV testing. However, there are concerns about the comparability and acceptability of self-sampling kits.

The main objective of this study is to compare the test characteristics of the human papillomavirus (HPV) self-sampling kit versus clinician-sampled HPV testing for cervical cancer screening. Potential participants will be identified from the Penn State Family and Community Medicine and OBGYN clinics after it is determined that they have abnormal findings on their (clinician-sampled) Pap/HPV test and require a follow-up colposcopy. The patient will be pre-screened by a study team member. If they are found to be eligible, a study team member will invite them to participate in the study.

After a participant enrolls in the study, a self-sampling kit is mailed to their home along with a Summary Explanation of Research consent form and instructional sheet. Participants will be asked to complete the kit two weeks before or after their colposcopy, giving them a 28 day collection window. Study team members will perform a follow-up survey after the sample is collected and provide reminder phone calls if needed.

ELIGIBILITY:
Inclusion Criteria:

* Penn State Health Patient
* Has an intact cervix
* Found to have abnormal findings on Pap/HPV test that requires a colposcopy
* Speaks, read, or writes well in English or Spanish

Exclusion Criteria:

* Pregnant
* Cognitively impaired
* Incarcerated
* Complete hysterectomy
* History of cervical treatment for abnormal Pap/HPV test (i.e. cryotherapy, loop electrosurgical excision procedure (LEEP))

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Moss, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Jennifer Moss, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Shieh Y, Eklund M, Sawaya GF, Black WC, Kramer BS, Esserman LJ. Population-based screening for cancer: hope and hype. Nat Rev Clin Oncol. 2016 Sep;13(9):550-65. doi: 10.1038/nrclinonc.2016.50. Epub 2016 Apr 13. PMID 27071351
- [Background] U. S. Preventive Services Task Force. Final recommendation statement: Cervical cancer: Screening; 2018. https://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatementFinal/cervical-cancer-screening2. Accessed 2018.
- [Background] Saslow D, Solomon D, Lawson HW, Killackey M, Kulasingam SL, Cain J, Garcia FA, Moriarty AT, Waxman AG, Wilbur DC, Wentzensen N, Downs LS Jr, Spitzer M, Moscicki AB, Franco EL, Stoler MH, Schiffman M, Castle PE, Myers ER; ACS-ASCCP-ASCP Cervical Cancer Guideline Committee. American Cancer Society, American Society for Colposcopy and Cervical Pathology, and American Society for Clinical Pathology screening guidelines for the prevention and early detection of cervical cancer. CA Cancer J Clin. 2012 May-Jun;62(3):147-72. doi: 10.3322/caac.21139. Epub 2012 Mar 14. PMID 22422631
- [Derived] Wong A, Morgis R, Entenman J, Ramirez SI, Hays AL, Wright TS, Scartozzi CM, Ruffin MT, Moss JL. Exploratory Analysis of Concordance Between Clinician-Collected and Self-Sampled Human Papillomavirus Tests in a Small Cohort of Average- and High-Risk Patients. Womens Health Rep (New Rochelle). 2024 Mar 13;5(1):259-266. doi: 10.1089/whr.2024.0004. eCollection 2024. PMID 38516651

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: The participants in this study were scheduled for a colposcopy procedure due to abnormal findings during their recent standard-of-care, clinical-collected cervical cancer screening.
Period: Overall Study
Arm/Group | Participants
Started | 22
Completed | 12
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 12
annual household income [Count of Participants; unit: Participants]
  <$50,000 | 2
  $50,000 + | 9
  unknown/not reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Concordance of Screening Results of the Self-Sampling Kit Compared to Clinician-collected Samples
Description: The primary outcome of this study is to analyze the number of participants with concordance of screening results of the self-sampling kit compared to clinician-collected HPV test, Pap smear results, and colposcopy.
Time Frame: Within two weeks of their colposcopy exam.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 12
Participants | 8

2. Secondary Outcome: Number of Completed Self-Sampling Kits
Description: The number of participants provided a kit vs. those who completed the sample collection
Time Frame: Within two weeks of their colposcopy exam.
Population: Total number of participants who were provided with a self-sampling kit.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 22
Participants | 12

3. Secondary Outcome: Number of Participants Who Reported Problems Using Self-Sampling Kits
Description: The number of participants, among those who completed the sample collection, who reported problems using the self-sampling kit.
Time Frame: Within two weeks of their colposcopy exam
Population: Total number of participants who returned the self-sampling kit.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event information was collected during the time between the clinician and self-sampled tests for all participants, which was 212 days or just over 7 months.
Groups:
- Participants: Participants were those scheduled for a colposcopy procedure due to abnormal findings during their recent standard-of-care, clinical-collected cervical cancer screening.
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
small sample size due to slow participant accrual, exclusion of patients who do not engage in health care (group most likely to benefit from self-sampling)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT04585243/Prot_SAP_002.pdf
  • Informed Consent Form (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04585243/ICF_003.pdf